CLINICAL TRIAL: NCT02385942
Title: KT-SNUBH U-health Cooperative Research: Target Selection and Consumers' Intention Research for Commercialization of the Pressure Ulcer Management u-Health Solution
Brief Title: KT(KT Corporation)-SNUBH(Seoul National University Bundang Hospital) U-health Cooperative Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chan-Yeong Heo (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Sponsor-Investigator, Chan-Yeong Heo, Assistant professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E-1206/158-001
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Pressure Ulcer
Keywords: u-health; chronic wound management; pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tele-consultation system (Other): compare the Live assessed wound size with the transmitted Smart phone-based wound size through Tele-consultation system
  Interventions: Device: Smart phone

INTERVENTIONS:
Device: Smart phone — * measure the Live assessed wound size and the transmitted Smart phone-based wound size
  * determine dressing materials using Smart phone-based tele-consultation

SUMMARY:
The purpose of this study is to analyse utility and compatibility of U-health solution service based on mobile for chronic wound management.

DETAILED DESCRIPTION:
In this study, 'the management of pressure ulcer' defined as procedures comprising wound assessment, wound dressing and infection control, visually evaluated the outcomes of 'the management of pressure ulcer' through the tele-consultation.

This study designed to draw service targets based on utility and compatibility of U-health solution service and to analyse whether health providers use U-health solution service.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has pressure ulcer or Health care provider for wound management

Exclusion Criteria:

* Subject who have Osteomyelitis
* Subject who have suppuration
* Subject who participated in other clinical trial within 30 days from screening date

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
concordance rate of wound size between live assessed wound size and transmitted wound size | a week from post treatment

SECONDARY OUTCOMES:
concordance rate of wound size between live assessed wound size and transmitted wound size | 2 weeks from post treatment
concordance rate of wound size between live assessed wound size and transmitted wound size | 3 weeks from post treatment
concordance rate of wound size between live assessed wound size and transmitted wound size | 4 weeks from post treatment

OTHER OUTCOMES:
Satisfaction degree of the tele-consultation as measured by questionnaire. | 4 weeks from post treatment
Usability survey | 4 weeks from post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea